CLINICAL TRIAL: NCT02842177
Title: Classic vs. Uterine Sound-sparing Approach for Insertion of Copper T380A Intrauterine Device
Brief Title: Evaluation of a Novel Technique for Intrauterine Contraceptive Devices Insertion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammed Khairy Ali, Dr, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NIUD
Record Dates: First submitted 2016-07-15; First posted 2016-07-22 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2017-03

CONDITIONS: Contraception

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group I (classic method) (Active Comparator)
  Interventions: Procedure: Classic group; Device: Cu-IUD
- uterine sound sparing group (Active Comparator)
  Interventions: Procedure: Classic group; Procedure: Uterine sounding sparing group; Radiation: Transvaginal ultrasound; Device: Cu-IUD

INTERVENTIONS:
Procedure: Classic group — The speculum was placed into the vagina and the cervix was cleansed with povidone iodine. After placement of single toothed vulsellum on the anterior lip of the cervix, for traction and fixation of the uterus, the uterine sound was inserted for determination of uterine length and uterine position followed by Cu-IUD insertion. The duration of IUD insertion were reported.
Procedure: Uterine sounding sparing group — after bimanual examination, the same sonographer (Level II experience) performed transvaginal /US using a SonoAce X6 machine (Medison, Korea) with transvaginal probe (4-8 MHz frequency, using an average 6.5 MHz). Firstly, he evaluated the uterine position. Then, he measured the endometrial and cervical stripe lengths in the sagittal view of the uterus and summed to have the actual length of the uterus; by which the IUD tube was adjusted before insertion.The same speculum and vulsellum were used and the IUD was inserted directly into the uterine cavity.
  Arms: uterine sound sparing group
Radiation: Transvaginal ultrasound
  Arms: uterine sound sparing group
Device: Cu-IUD

SUMMARY:
The intrauterine devices are a safe, reliable, long-acting and reversible contraceptive method. It is also sound safe and cheap contraceptive methods available and is nearly maintenance free for up to 10 years.

The fear and the pain associated with intrauterine devices insertion consider barriers to using this contraception method, this is because that the mucosal lining of female genital tract is highly sensitive to touch and pain. However; most of small procedures done in this sensitive area are performed without analgesia.

The pain during intrauterine devices insertion is due to application of the tenaculum , traction of the cervical canal, passing the uterine sound, insertion of the intrauterine devices through the cervix, and irritation of the endometrial lining by the intrauterine devices .

Previous studies have reported different lines to decrease pain during intrauterine device insertion starting by simple methods such as pre-insertion ibuprofen use, intracervical or intrauterine lidocaine and misoprostol up to paracervical blocks.

Previous studies, in literature, have found that the most painful steps during intrauterine devices insertion were uterine sounding then intrauterine device insertion itself, followed by tenaculum placement. One recent study addressed pain effect using an atraumatic vulsellum and a single-tooth tenaculum on pain perception during intrauterine devices and found no difference in reported pain.

ELIGIBILITY:
Inclusion Criteria:

* Women requesting intrauterine contraceptive device as a contraction

Exclusion Criteria:

* Uterine abnormalities
* Endometrial lesions,
* Adenomyosis
* Fibroids
* Intrauterine adhesions.
* Chronic pelvic pain
* Spasmodic dysmenorrhea
* History of cervical surgery

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 92 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Successful intrauterine device insertion | 5 minutes
  defined by a distance from the intrauterine device to the end of endometrial line of less than 25 mm The degree of total pain perception during intrauterine contraceptive insertion measured by visual analogue scale

SECONDARY OUTCOMES:
The degree of pain during intrauterine device insertion | 5 minutes
  measured by Visual Analog Pain Scale
the duration of intrauterine device insertion | 5 minutes
  The time between start of IUD insertion and the end of the procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Women Health Hospital - Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Yes